CLINICAL TRIAL: NCT01027260
Title: A Randomized, Placebo Controlled Study on the Efficacy of Itopride HCI on Irritable Bowel in Patients of Irritable Bowel Syndrome With Constipation (IBS-C)
Brief Title: Study to Evaluate the Role of Itopride HCI in Patients With Irritable Bowel Syndrome With Predominant Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R10-257
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Itopride 50 mg (Active Comparator)
  Interventions: Drug: Itopride HCI 50 mg
- Itopride 100 mg (Active Comparator)
  Interventions: Drug: Itopride HCI 100 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itopride HCI 50 mg — Variable dosing
  Other Names: ABT-654; Itopride HCI; Ganaton
  Arms: Itopride 50 mg
Drug: Itopride HCI 100 mg — Variable dosing
  Other Names: ABT-654; Itopride HCI; Ganaton
  Arms: Itopride 100 mg
Drug: Placebo — Variable dosing
  Arms: Placebo

SUMMARY:
Patients suffering from Irritable Bowel Syndrome with predominant constipation will be provided with the study medication. The study medication will be evaluated for its efficacy in relieving the symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient fulfilling the Rome III criteria for IBS-C
2. Signed informed consent at screening visit

Exclusion Criteria:

1. Patients having significant diarrhea at least 25% of the time during the past 3 months
2. Patients having alarm symptoms or signs
3. Chronic diarrhea
4. History of gastrointestinal haemorrhage, mechanical obstruction or perforation
5. Patient with clinically relevant ECG abnormalities (prolonged QT interval)
6. Active psychiatric disorder that would interfere with the study objectives
7. Health conditions (e.g. age related impairment of cognitive functions) that would interfere with the study objectives or might impair the compliance of the patient
8. Severe hepatic, renal, cardiac, metabolic, haematological or malignant diseases (including prolactin dependent tumours) or clinically relevant deviations in laboratory values (AST/ALT greater than twice the upper limit of normal, serum creatinine * 2 mg/dl [177 µmol/l] according to the medical judgement of the investigator
9. Patient with hypokalemia (serum potassium < 3.5 mmol/l).
10. History of any known hypersensitivity to the ingredients of the investigational drug
11. Pregnancy or lactation
12. Women with childbearing potential who do not apply a medically accepted method of contraception.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 268 (Actual)
Dates: Start 2008-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Patients will be asked a simple but well validated question "If there is a satisfactory relief of the symptoms" | 2 weeks and 4 weeks after the start of the treatment

SECONDARY OUTCOMES:
Subjects will be assessed based on Irritable Bowel Syndrome Severity Score (IBSSS). | 2 weeks and 4 weeks after the start of the treatment
Safety based on the laboratory tests before and at the end of the treatment. | 4 weeks during the treatment period and 4 weeks following post- therapy period.

CONTACTS AND LOCATIONS:
Locations (4):
- Pakistan (4):
  - Site Reference ID/Investigator# 5870, Karachi
  - Site Reference ID/Investigator# 21441, Karachi
  - Site Reference ID/Investigator# 6130, Lahore
  - Site Reference ID/Investigator# 8535, Rawalpindi